CLINICAL TRIAL: NCT06744920
Title: A Randomized, Double-blind, Placebo-controlled Phase III Study to Evaluate the Efficacy, Safety, and Tolerability of Remibrutinib in Patients With Generalized Myasthenia Gravis, Followed by an Open-label Extension Phase
Brief Title: A Study to Investigate the Efficacy, Safety and Tolerability of Remibrutinib Versus Placebo in Adult Patients With Generalized Myasthenia Gravis
Acronym: RELIEVE
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLOU064O12301; 2023-510026-32 (Other: EU CTIS)
Record Dates: First submitted 2024-12-17; First posted 2024-12-20 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Generalized Myasthenia Gravis
Keywords: Myasthenia Gravis; gMG; Generalized Myasthenia Gravis; LOU064; Remibrutinib; placebo-controlled; double-blind; phase III
MeSH Terms: conditions — Myasthenia Gravis | interventions — remibrutinib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Remibrutinib arm (Experimental): Core Part: Remibrutinib tablet taken orally
  [Extension Part: Open-label remibrutinib tablet taken orally]
  Interventions: Drug: Remibrutinib (Blinded); Drug: Remibrutinib (Open Label)
- Placebo arm (Placebo Comparator): Core Part: Placebo tablet taken orally
  [Extension Part: Open-label remibrutinib tablet taken orally]
  Interventions: Other: Placebo; Drug: Remibrutinib (Open Label)

INTERVENTIONS:
Drug: Remibrutinib (Blinded) — Remibrutinib (Blinded) active treatment
  Other Names: LOU64
  Arms: Remibrutinib arm
Other: Placebo — Placebo
  Arms: Placebo arm
Drug: Remibrutinib (Open Label) — Remibrutinib (Open Label) active treatment
  Other Names: LOU064

SUMMARY:
A study to evaluate the efficacy, safety and tolerability of Remibrutinib versus placebo in adult patients with Generalized Myasthenia Gravis who are on stable, standard-of-care (SOC) treatment.

DETAILED DESCRIPTION:
This study is a randomized, double-blind, placebo-controlled, multicenter, Phase III study, to evaluate the efficacy, safety and tolerability of remibrutinib in gMG patients who are on stable SOC treatment. Approximately 180 eligible participants will be randomized in a ratio of 1:1, to receive either remibrutinib or matching placebo.

The study consists of a Core Part (6-months double-blind treatment) and an Extension Part (up to 60-month open-label treatment).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with gMG (age 18-75 years)
* Confirmed diagnosis of Myasthenia Gravis Foundation of America (MGFA) Class II-IV gMG at screening and likely not in need of a respirator for the duration of the study, as judged by the Investigator
* Documented evidence of positive serologic testing for AChR+ antibody or MuSK+ antibody at screening, OR seronegative for both AChR and MuSK antibodies at screening
* Baseline MG-ADL score ≥ 6 with ≥ 50% of the total score due to non ocular symptoms
* Participants who have been on a stable dose of standard-of-care treatment as specified in the protocol
* Able to safely swallow the study medication according to investigator clinical judgement based on a bedside swallowing test or another formal swallowing test in line with local practice, both at Screening and Baseline

Exclusion Criteria:

* Prior to baseline have been treated with intravenous immunoglobulins or plasma exchange (IVIg/PLEX) in the past month, with rituximab in the past 6 months, eculizumab in the past 2 months, ravulizumab or other complement inhibitors in the past 3 months, efgartigimod or other anti-FcRn therapies in the past 3 months, or had a thymectomy in the past 6 months or a planned thymectomy during the trial period
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception during dosing and for 1 week after stopping of study treatment

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-02-07 (Actual); Primary Completion 2028-02-27 (Estimated); Study Completion 2033-02-26 (Estimated)

PRIMARY OUTCOMES:
Change from baseline to Month 6 in Myasthenia Gravis Activity of Daily Living (MG-ADL) total score | Baseline to Month 6
  The MG-ADL is a categorical scale that assesses MG symptoms and their effects on daily activities. MG-ADL is composed of items related to patient's assessment of functional disability secondary to ocular (2 items), bulbar (3 items), respiratory (1 item), and gross motor or limb (2 items) impairment related to effects from MG.
  Each item is assessed on a 4-points scale where a score 0 represents normal function and a score 3 represents loss of ability to perform that function (total score 0 to 24).

SECONDARY OUTCOMES:
Change from baseline to Month 6 in Quantitative Myasthenia Gravis (QMG) total score | Baseline to Month 6
  The Quantitative Myasthenia Gravis (QMG) Score is a 13-item direct physician assessment scoring system that quantifies disease severity, based on impairments of body functions and structures. The total QMG score ranges from 0 to 39, where higher scores indicated greater disease severity. The QMG score is composed of the following items: ocular (2 items), facial (1 item), bulbar (2 items), gross motor (6 items), axial (1 item) and respiratory (1 item).
Proportion of participants with ≥ 5 points reduction from baseline to Month 6 of QMG total score without rescue medication and/or strongly confounding prohibited medication | Baseline to Month 6
  The Quantitative Myasthenia Gravis (QMG) Score is a 13-item direct physician assessment scoring system that quantifies disease severity, based on impairments of body functions and structures. The total QMG score ranges from 0 to 39, where higher scores indicated greater disease severity. The QMG score is composed of the following items: ocular (2 items), facial (1 item), bulbar (2 items), gross motor (6 items), axial (1 item) and respiratory (1 item).
Proportion of participants with ≥ 3 points reduction from baseline to Month 6 of Myasthenia Gravis Activity of Daily Living (MG-ADL) scale total score without rescue medication and/or strongly confounding prohibited medication | Baseline to Month 6
  The MG-ADL is a categorical scale that assesses MG symptoms and their effects on daily activities. MG-ADL is composed of items related to patient's assessment of functional disability secondary to ocular (2 items), bulbar (3 items), respiratory (1 item), and gross motor or limb (2 items) impairment related to effects from MG.
  Each item is assessed on a 4-points scale where a score 0 represents normal function and a score 3 represents loss of ability to perform that function (total score 0 to 24).
Proportion of participants achieving Minimal Symptom Expression (MSE) at Month 6, defined as MG-ADL score of 0 or 1 at Month 6 without rescue therapy and/or strongly confounding prohibited medication | Month 6
  The MG-ADL is a categorical scale that assesses MG symptoms and their effects on daily activities. MG-ADL is composed of items related to patient's assessment of functional disability secondary to ocular (2 items), bulbar (3 items), respiratory (1 item), and gross motor or limb (2 items) impairment related to effects from MG.
  Each item is assessed on a 4-points scale where a score 0 represents normal function and a score 3 represents loss of ability to perform that function (total score 0 to 24).
Change from baseline to Month 6 in Myasthenia Gravis Composite score (MGC) total score | Baseline to Month 6
  The MGC is a 10-item instrument that measures the symptoms and signs of MG based on physician examination and patient history. Items relate to ptosis, double vision, eye closure, talking, chewing, swallowing, breathing, neck flexion, shoulder abduction, and hip flexion. Each item is scored on an ordinal scale with 4 possible categories and weighted. The total score ranges from 0 to 50, where higher scores indicating more severe impairments.
Change from baseline to Month 6 in revised Myasthenia Gravis Quality of Life Questionnaire (MG-QOL15r) survey score | Baseline to Month 6
  The revised MG-QoL15 is a 15-item health related quality of life questionnaire completed by participants, designed to measure quality of life in gMG. Items on the MG-QoL15 relate to physical, social, and psychological components and are scored from 0 (not at all) to 2 (very much). The cumulative scores range from 0 to 30, with higher scores representing worse quality of life and dissatisfaction with MG-related dysfunction.
Incidence of adverse events | Baseline to Month 6
  Incidence of adverse events including changes in clinical laboratory values, vital signs, electrocardiograms and suicidality results qualifying and reported as AEs.
Proportion of time during which participants showed a reduction of ≥ 2 points in MG-ADL total score, that was maintained up to Month 6 | Baseline to Month 6
  The MG-ADL is a categorical scale that assesses MG symptoms and their effects on daily activities. MG-ADL is composed of items related to patient's assessment of functional disability secondary to ocular (2 items), bulbar (3 items), respiratory (1 item), and gross motor or limb (2 items) impairment related to effects from MG. Each item is assessed on a 4-points scale where a score 0 represents normal function and a score 3 represents loss of ability to perform that function (total score 0 to 24).
Proportion of early MG-ADL responders during treatment (early responders with first MG-ADL improvement from baseline of ≥ 2 points occurring by week 4） | Baseline to week 4
  The MG-ADL is a categorical scale that assesses MG symptoms and their effects on daily activities. MG-ADL is composed of items related to patient's assessment of functional disability secondary to ocular (2 items), bulbar (3 items), respiratory (1 item), and gross motor or limb (2 items) impairment related to effects from MG. Each item is assessed on a 4-points scale where a score 0 represents normal function and a score 3 represents loss of ability to perform that function (total score 0 to 24). Participants with a first MG-ADL improvement from baseline of ≥ 2 points occurring by week 4 are considered early responders.
Change from baseline to Month 6 in EuroQol-5 Dimensions-5 Level (EQ-5D-5L) | Baseline to Month 6
  The EQ-5D-5L is a widely used questionnaire designed to assess health status in adults. The measure is divided into two distinct sections, the descriptive system and the EQ visual analogue scale (EQ VAS). The first section includes one item addressing each of five dimensions (mobility, self-care, usual activity, pain/discomfort, and anxiety/depression). Participants rate each of these items from 1 of the 5 levels: no problems, slight problems, moderate problems, severe problems, or unable to/extreme. A composite health state is then defined by combining the levels for each dimension into a 5-digit number. The second section includes the EQ visual analogue scale (EQ VAS) that measures self-rated (global) health status utilizing a vertically oriented visual analogue scale where 100 represents the "best imaginable health state" and 0 represents the "worst imaginable health state." Respondents are asked to rate their current health by placing a mark along this continuum.
Proportion of participants achieving a reduction from baseline of ≥ 3 points in MGC total score at Month 6 | Baseline to Month 6
  The MGC is a 10-item instrument that measures the symptoms and signs of MG based on physician examination and patient history. Items relate to ptosis, double vision, eye closure, talking, chewing, swallowing, breathing, neck flexion, shoulder abduction, and hip flexion. Each item is scored on an ordinal scale with 4 possible categories and weighted. The total score ranges from 0 to 50, where higher scores indicating more severe impairments.
Change from baseline in MG-ADL total score | Baseline to Month 66
  The MG-ADL is a categorical scale that assesses MG symptoms and their effects on daily activities. MG-ADL is composed of items related to patient's assessment of functional disability secondary to ocular (2 items), bulbar (3 items), respiratory (1 item), and gross motor or limb (2 items) impairment related to effects from MG. Each item is assessed on a 4-points scale where a score 0 represents normal function and a score 3 represents loss of ability to perform that function (total score 0 to 24).
Proportion of participants achieving a reduction from core part in oral corticosteroids (OCS) dose till the end of extension part | Baseline to month 66
  Participants receiving oral corticosteroids are required to be on a stable dose for at least 4 weeks prior to baseline. The dose can be reduced or discontinued during the open label extension period at investigator discretion. Oral corticosteroids use will be recorded.
Incidence of adverse events | Month 7 to month 66
  Incidence of adverse events including changes in clinical laboratory values, vital signs, electrocardiograms and suicidality results qualifying and reported as AEs.

CONTACTS AND LOCATIONS:
Locations (80):
- United States (18):
  - Neuromuscular Research Center, Phoenix, Arizona
  - Honor Health Research Institute, Scottsdale, Arizona
  - Fullerton Neuro and Headache Ctr, Fullerton, California
  - University Of Southern California, Los Angeles, California
  - Univ Cali Irvine ALS Neuromuscular, Orange, California
  - SFM Clinical Research LLC, Boca Raton, Florida
  - Homestead Assoc In Research Inc, Homestead, Florida
  - AdventHealth, Orlando, Florida
  - Neurological Services of Orlando PA, Orlando, Florida
  - Mid Atlantic Epilepsy and Sleep Ctr, Bethesda, Maryland
  - Michigan State University-Department of Neurology, East Lansing, Michigan
  - Dent Neurological Institute, Buffalo, New York
  - Univ of Cincinnati Medical Center, Cincinnati, Ohio
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Houston Methodist Hospital, Houston, Texas
  - UT Health Science Center, Houston, Texas
  - University of WA Division of Cardio, Seattle, Washington
  - Center for Neurological Disorders G, Greenfield, Wisconsin
- Novartis Investigative Site, Rosario, Santa Fe Province, Argentina
- Australia (3):
  - Novartis Investigative Site, Kogarah, New South Wales
  - Novartis Investigative Site, Fitzroy, Victoria
  - Novartis Investigative Site, Southport
- Novartis Investigative Site, Leuven, Vlaams Brabant, Belgium
- Canada (2):
  - Novartis Investigative Site, London, Ontario
  - Novartis Investigative Site, Ottawa, Ontario
- China (6):
  - Novartis Investigative Site, Guangzhou, Guangdong
  - Novartis Investigative Site, Shijiazhuang, Hebei
  - Novartis Investigative Site, Wuhan, Hubei
  - Novartis Investigative Site, Wuxi, Jiangsu
  - Novartis Investigative Site, Changchun, Jilin
  - Novartis Investigative Site, Shanghai
- France (4):
  - Novartis Investigative Site, Bordeaux
  - Novartis Investigative Site, Nice
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Toulouse
- Georgia (2):
  - Novartis Investigative Site, Kutaisi
  - Novartis Investigative Site, Tbilisi
- India (6):
  - Novartis Investigative Site, Mangalore, Karnataka
  - Novartis Investigative Site, Nashik, Maharashtra
  - Novartis Investigative Site, New Delhi, National Capital Territory of Delhi
  - Novartis Investigative Site, Ludhiana, Punjab
  - Novartis Investigative Site, Vellore, Tamil Nadu
  - Novartis Investigative Site, Hyderabad, Telangana
- Novartis Investigative Site, Bergamo, BG, Italy
- Japan (11):
  - Novartis Investigative Site, Sapporo, Hokkaido
  - Novartis Investigative Site, Nishinomiya, Hyōgo
  - Novartis Investigative Site, Hanamaki, Iwate
  - Novartis Investigative Site, Sendai, Miyagi
  - Novartis Investigative Site, Suita, Osaka
  - Novartis Investigative Site, Higashi-Matsuyama, Saitama
  - Novartis Investigative Site, Koshigaya, Saitama
  - Novartis Investigative Site, Shinjuku Ku, Tokyo
  - Novartis Investigative Site, Chiba
  - Novartis Investigative Site, Fukushima
  - Novartis Investigative Site, Hiroshima
- Poland (10):
  - Novartis Investigative Site, Lublin, Lublin Voivodeship
  - Novartis Investigative Site, Krakow, POL
  - Novartis Investigative Site, Bydgoszcz, Woj Kujawsko Pomorskie
  - Novartis Investigative Site, Bydgoszcz
  - Novartis Investigative Site, Katowice
  - Novartis Investigative Site, Lodz
  - Novartis Investigative Site, Lublin
  - Novartis Investigative Site, Poznan
  - Novartis Investigative Site, Skorzewo
  - Novartis Investigative Site, Warsaw
- Romania (3):
  - Novartis Investigative Site, Brasov
  - Novartis Investigative Site, Bucharest
  - Novartis Investigative Site, Sibiu
- South Korea (3):
  - Novartis Investigative Site, Seoul, Korea
  - Novartis Investigative Site, Busan
  - Novartis Investigative Site, Seoul
- Spain (5):
  - Novartis Investigative Site, L'Hospitalet de Llobregat, Barcelona
  - Novartis Investigative Site, Lleida
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Málaga
  - Novartis Investigative Site, Valencia
- Taiwan (4):
  - Novartis Investigative Site, Kaohsiung City
  - Novartis Investigative Site, Tainan
  - Novartis Investigative Site, Taipei
  - Novartis Investigative Site, Taoyuan District

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations. This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com.